CLINICAL TRIAL: NCT05045625
Title: Effects of Novel SCS Paddle on Intraoperative Neuromonitoring Recording
Brief Title: Intraoperative Neuromonitoring Recording With a Novel SCS Paddle
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Albany Medical College (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: Microleads 5151
Record Dates: First submitted 2021-09-07; First posted 2021-09-16 (Actual); Results first posted 2023-01-12 (Actual); Last update posted 2023-03-01 (Actual); Status verified 2023-02

CONDITIONS: Chronic Pain; Neuropathic Pain; Failed Back Surgery Syndrome; Complex Regional Pain Syndromes
Keywords: Spinal cord stimulation; chronic pain
MeSH Terms: conditions — Chronic Pain; Neuralgia; Failed Back Surgery Syndrome; Complex Regional Pain Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Study Group (Experimental): Twelve patients offered SCS for standard of care were also invited to participate in this study, in which a study electrode was temporarily placed intraoperatively and neuromonitoring was done per our routine standard-of-care
  Interventions: Device: HD Study Electrode

INTERVENTIONS:
Device: HD Study Electrode — The HD Study Electrode is an array of 8 columns of stimulation contacts arranged in 8 rows with a low-volume electrode body. This array of stimulation electrodes contact patterns of bi-poles and tri-poles may be applied to the spinal cord for assessment of dermatomal selective stimulation patterns.

SUMMARY:
The purpose of this study is to demonstrate safety and efficacy of a new spinal cord stimulation paddle electrode which is able to target the dorsal horns, dorsal nerve roots, and dorsal columns. The research electrode ("Study Electrode") is designed to answer basic physiological clinical research questions. It may inform future device therapy development, but the Study Electrode is not a product that will be marketed or sold. The Investigators believe the protocol is a Non-Significant Risk study answering basic physiological research questions, which may be performed under hospital IRB approval.

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing a spinal cord stimulation procedure for neuropathic pain
* must be fluent in English as well as mentally competent to read and answer the questionnaires, as well as complete pain assessment exams.
* subjects must be able to give informed consent.

Exclusion Criteria:

* patients who are not undergoing thoracic spinal cord stimulation for chronic neuropathic pain

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2020-01-10 (Actual); Primary Completion 2021-03-20 (Actual); Study Completion 2021-03-20 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Albany Medical College, Albany, New York, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Study Group
Started | 12
Completed | 9
Not Completed | 3
Not completed — Lost to Follow-up | 3

BASELINE CHARACTERISTICS:
Arm/Group | Study Group
Number analyzed (Participants) | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.75 (14.75)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 11
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 12
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Numeric Rating Scale (NRS)
Description: Patients rate their pain on a scale from 0-10; 0 being not in pain and 10 being worst pain imaginable. A higher score indicates worse outcome.
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Study Group
Number analyzed (Participants) | 9
score on a scale | 5.333333333 (2.115700942)

2. Secondary Outcome: McGill Pain Questionnaire (MPQ)
Description: Patients select words that describe their pain. There are a total of 15 words. A higher score (more words selected) indicates worse outcome with a range from 0-15.
Time Frame: 3 month
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Study Group
Number analyzed (Participants) | 9
score on a scale | 8.222222222 (2.886751346)

3. Secondary Outcome: Oswestry Disability Index (ODI)
Description: This is a multiple choice style scale where patients are presented with an activity and asked to select a description which best matches their ability to perform that activity. Multiple choice options are then scored on a scale from 0-5; where 0 is no issues performing the activity and 5 is cannot perform activity. A higher score indicates worse outcome. The range in scores is from 0-100.
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Study Group
Number analyzed (Participants) | 9
units on a scale | 50 (17.13086882)

4. Secondary Outcome: Pain Catastrophizing Scale (PCS)
Description: Patients are presented with a series of statements and they are asked to rate on a scale from 0-4, how often these statements apply to them when they are in pain. 0= never and 4= always. A higher score indicates worse outcome. Scores range from 0-52.
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Study Group
Number analyzed (Participants) | 9
units on a scale | 18 (12.43267584)

5. Secondary Outcome: Beck Depression Index (BDI)
Description: This is a multiple choice style scale where patients are asked to select a statement related to a feeling of sadness or a component of depression. Multiple choice options are then scored on a scale from 0-3; where 0 is they do not feel that way and 3 is they do feel that way. A higher score indicates worse outcome. Scores range from 0-63
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Study Group
Number analyzed (Participants) | 9
units on a scale | 14.33333333 (12.35198075)

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Study Group
All-Cause Mortality (participants affected / at risk) | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12
Other Adverse Events (participants affected / at risk) | 1/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Study Group (N=12)
intraoperative (Surgical and medical procedures) | 1 (1) — During optimization of lead placement, we noticed that one contact of the 64 became dislodged. We were able to retrieve it easily with suction.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2021-07-02): https://cdn.clinicaltrials.gov/large-docs/25/NCT05045625/Prot_SAP_ICF_000.pdf